CLINICAL TRIAL: NCT03569150
Title: Culturally-Adapting a Communication Intervention to Improve End-of-Life Palliative Care Health Literacy on Two Native American Reservations: An Academic-Tribal Partnership
Brief Title: Culturally-Adapting a Communication Intervention to Improve Palliative Care Literacy on Two Native American Reservations
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not funded.
Sponsor: South Dakota State University (Other)
Collaborators: Southcentral Foundation (Other); Indian Health Service (IHS) (U.S. Federal Agency); Rosebud Sioux Tribe Health Administration (Unknown); Oglala Sioux Tribe Health Administration (Unknown); California State University, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SDSU4909
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Advance Care Planning
Keywords: palliative care; end-of-life care; advance care planning; communication; health literacy; serious life-limiting illness
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: cluster-assigned pilot, wait-list control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Rosebud) (Other): The intervention is: Native Americans patients with a serious life-limiting illness will have an advance care planning discussion with an interdisciplinary healthcare professional trained in the culturally-adapted COMFORT Communication Curriculum.
  Interventions: Other: Cultural adaptation/implementation COMFORT CC
- Control (Pine Ridge) (No Intervention): In the control group, Native American patients with a serious life-limiting illness will receive usual care. The healthcare professionals have not undergone training in the culturally-adapted COMFORT Communication Curriculum.

INTERVENTIONS:
Other: Cultural adaptation/implementation COMFORT CC — The COMFORT Communication Curriculum (CC) will be culturally-adapted for 2 Native American reservation communities. The investigators will then implement the culturally-adapted COMFORT Communication Curriculum in 2 tribal communities by training interdisciplinary healthcare professionals to conduct culturally-respectful and relevant Advance Care Planning. The investigators will then conduct a cluster-assigned pilot, wait-list controlled trial of the culturally-adapted COMFORT Communication Curriculum in 2 tribal communities to evaluate feasibility, acceptability, and perceived effectiveness by comparing 30 Native Americans completing Advance Care Planning with a trained healthcare professional and 30 Native Americans receiving usual care.
  Arms: Intervention (Rosebud)

SUMMARY:
This study will evaluate the feasibility, acceptability, and perceived effectiveness of the culturally-adapted COMFORT Communication Curriculum in two Native American reservation communities. Participants in one community will have an advance care planning conversation with a healthcare professional trained in the the culturally-adapted curriculum. Participants in the other community will receive usual care.

DETAILED DESCRIPTION:
Advance care planning (ACP) is an important component of palliative care (PC), and is a critical, ongoing dialogue between health care professionals (HCPs), patients, and families; where patients' comprehension of their illness and illness progression, goals of care, and treatment choices are discussed. Essential to ACP is the interdisciplinary team, where each member must be comfortable and confident initiating conversations about quality of life and end-of-life (EOL) care. ACP is often hindered by low health literacy, including PC health literacy, uncertainty regarding illness trajectory and end-of-life palliative care (EOLPC) options, and lack of awareness about ACP among patients. For HCPs, discomfort, lack of EOL communication training, and knowledge of cultural differences are often barriers to ACP. Foundational to ACP is PC health literacy, which necessitates considering semantics, eliminating misconceptions, and recognizing uncertainty. Ensuring access to ACP for patients with serious life-limiting illness requires that all healthcare disciplines receive evidence-based EOLPC communication training. The COMFORT communication curriculum (CC) is an intervention that trains interdisciplinary HCPs to provide patient- and family-centered EOLPC communication. Patient outcomes related to this intervention have not been studied. Moreover, the curriculum's efficacy and fit has not been specifically tested with minority groups. Native Americans (NA) are disproportionately affected by serious life-limiting conditions and life expectancy is 4 years less than all other US races. Despite greater morbidity and mortality, NAs use of PC is largely unknown. Yet, it has been identified that tribal communities are requesting EOLPC services and will participate in ACP when conducted in a culturally-respectful manner. There is an urgent need to develop culturally-relevant communication approaches specific to EOLPC, including ACP, for use with NAs with serious life-limiting illness. The investigators propose a collaborative clinical trial to: 1) Culturally-adapt the COMFORT CC for pilot testing with NA communities; 2) Implement the culturally-adapted COMFORT CC in 2 tribal communities by training 20 interdisciplinary (nurses, social workers, primary care providers) HCPs to conduct culturally-respectful and relevant ACP; 3) Conduct a pilot, wait-list controlled trial of the culturally-adapted COMFORT CC in 2 tribal communities to evaluate feasibility, acceptability, and perceived effectiveness by comparing 30 NAs completing ACP with a trained HCP and 30 NAs receiving usual care. Implementing a culturally-relevant communication intervention to improve EOLPC health literacy is a high priority for the Rosebud and Pine Ridge reservations in South Dakota. This proposed study will culturally-adapt and evaluate the COMFORT CC on these 2 reservations and will provide the foundation for an R01-funded intervention study that could positively impact EOLPC literacy and outcomes among the 566 US federally recognized NA tribes.

ELIGIBILITY:
Inclusion Criteria:

Focus Groups. Aim 1.1: Patient eligibility criteria: 1) Native American; 2) 18 years old or greater; 3) and diagnosis with one or more serious life-limiting illness, such as renal failure, cancer, or heart disease, as defined by the International Statistical Classification of Diseases and Related Health Problems (ICD-10). Caregiver eligibility criteria: 1) 18 years old or greater; 2) primary caregiver of a family member participant. Healthcare Professional eligibility: employment 1 year or more as a nurse, social worker, or primary care provider at Indian Health Service. An Elder is eligible if he/she is Native American and an identified elder in the community. Tribal health leader/representative inclusion criteria: 1) Native American; 2) 18 years old or greater; 3) live in the community; 4) employed by tribal health administration.

Cognitive Interviews. Aim 1.2: The investigators will recontact and reconsent those patients, family caregivers, and Elders who participated in the focus groups (Aim 1.1) (Total of 10; 5 per site) to conduct interviews assessing the culturally-adapted COMFORT Communication Curriculum's cultural relevance and fit.

COMFORT Communication Curriculum Training. Aim 2.1: Healthcare Professionals (nurses, social workers, primary care providers) will be recruited through Indian Health Service nursing and clinic administrators and must be employed for 1 year or more by Rosebud Indian Health Service to participate in the COMFORT Communication Curriculum education (Total of 10). The wait-list control arm (Pine Ridge Healthcare Professionals; total of 10) will receive the education following completion of data collection in the intervention group. Participants will be recruited through Indian Health Service nursing and clinic administrators and must be employed for 1 year or more by Pine Ridge Indian Health Service to participate in the COMFORT Communication Curriculum education.

Cluster-assigned wait-list control Trial. Aims 3.1 and 3.2: The intervention will be applied to Rosebud; Pine Ridge will serve as the control community. We will recruit patients (Total of 30) to the intervention arm (Rosebud Indian Health Service) from the outpatient clinics. For Pine Ridge, the electronic health record will be used to identify 30 participants from the outpatient clinic meeting the same eligibility criteria (Native American, 18 years of age or greater, ICD-10 codes identifying serious life-limiting illness) as the Rosebud participants. Patient eligibility criteria are the same as Aim 1.1. Patient eligibility will be identified by trained project Indian Health Service personnel at both sites.

Cognitive Interviews. Aim 3.3: Participants from the intervention arm (Rosebud) who participated in Aim 3.1 and 3.2 (total of 10 of the 30) will be asked to participate in an interview regarding their Advance Care Planning. Interested participants will provide a contact phone number and be given an information sheet by trained project Indian Health Service personnel regarding the interview purpose. Researchers will contact the participant via phone within 2 business days of visit and if still agreeable, schedule a face-to-face interview within 14 business days of advance care planning, where they will be reconsented.

Exclusion Criteria:

* Participants not meeting the inclusion criteria for the above aims will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Documentation of advance care planning and advance directive completion | Project Year 02, Quarter 2 and Quarter 3
  The investigators will evaluate this outcome by measuring the presence or absence of advance care planning documentation and advance directive completion in the patient's electronic health record at both the intervention and control sites.

SECONDARY OUTCOMES:
Level of uncertainty perceived in illness | Project Year 02, Quarter 2 and Quarter 3
  This will be evaluated by patient report using the validated Mishel Uncertainty in Illness Scale- Community (MUIS-C) pre and post outpatient clinic visit only at the intervention site. Uncertainty in illness (construct) is often discussed in relationship to health literacy, and for purposes of this study, end of life palliative care health literacy. This outcome will be evaluated by patient report using the validated MUIS-C, which has been used extensively in cancer, cardiac, and chronic illness patients and in cross-cultural studies. The MUIS-C is a 23-item Likert-format scale, where patients score items from 1 (strongly disagree) to 5 (strongly agree). The total score range is 23-115, with higher scores indicating a greater level of uncertainty. Reported Cronbach's alphas are 0.74 to 0.92.
Patient satisfaction with the intervention | Project Year 02, Quarter 2 and Quarter 3
  The investigators will conduct cognitive interviews with patients that participated in the intervention and completed a MUIS-C, only with intervention participants.

OTHER OUTCOMES:
Healthcare Professional Comfort with Palliative and End-of-life Communication | Project Year 02, Quarter 1 and Quarter 2
  Healthcare professionals participating in the COMFORT Communication Curriculum (CC) training will complete a C-COPE (Comfort with Communication in Palliative and End of Life Care) questionnaire before and after training. This will be done only at the intervention site.The C-COPE operationalizes the key components within the COMFORT CC and is a 28-item instrument including 2-ranked items and 26 Likert-format items, where healthcare professionals score items from 1 (not difficult) to 5 (very difficult). The range of possible C-COPE total scores is 26-130, with higher scores indicating less comfort with end of life palliative care communication, while rated items are categorized according to patient, family, and team communication. Preliminary psychometric analysis of test-retest reliability with ICC > 0.77, internal reliability for total score with Cronbach's alpha = 0.91.

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Isaacson, PhD, Principal Investigator — South Dakota State University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available beginning 6 months and ending 5 years following article publication. Person(s) requesting data will complete a data request form.
Access Criteria: Data access requests will be reviewed first by an Independent Review Panel and if appropriate forwarded onto the tribal entities for final approval.